CLINICAL TRIAL: NCT01773564
Title: Comparison Between Two Types of Semipermeable Dressings of New Generation in the Prevention of Intravascular Catheters Related Complications in Intensive Care.
Brief Title: Comparison of Two New Generation Dressings in Intensive Care (ADVANCED)
Acronym: ADVANCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12SC03; 2012-A00734-39 (Other: ID RCB)
Record Dates: First submitted 2012-11-07; First posted 2013-01-23 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Complication of Catheter
Keywords: Dressings, Prevention,

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Available current hospital dressing (Active Comparator): Control group: depending on the type of dressing available at the hospital, either 3M™ HP Dressing or Smith & Nephew IV3000 ™
  Interventions: Device: Current hospital dressing
- 3M™ IV Advanced Securement dressing (Experimental): New generation transparent dressing
  Interventions: Device: 3M™ IV Advanced Securement dressing

INTERVENTIONS:
Device: Current hospital dressing — Patients were assigned to either arm following a randomization scheme 1:1.
  Other Names: 3M™ HP Dressing or Smith & Nephew IV3000 ™
  Arms: Available current hospital dressing
Device: 3M™ IV Advanced Securement dressing — Patients were assigned to either arm following a randomization scheme 1:1.
  Arms: 3M™ IV Advanced Securement dressing

SUMMARY:
Intravascular devices in intensive care units are often associated to complications. The investigators estimate that 23.5% of catheters placed and used in intensive care are subject to at least one complication; the investigators goal is to demonstrate the effectiveness of the new Tegaderm ™ IV Advanced dressings to achieve a decrease of 35% in the number of complications associated with intravascular catheters in intensive care.

DETAILED DESCRIPTION:
randomized controlled trial of 2 intravascular dressings in Intensive care unit

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with a central venous catheter, an arterial catheter, a hemodialysis catheter, a Swan Ganz catheter or a peripheral catheter inserted in the ICU or within the 24 before their arrival at the ICU in another ICU setting.
* Patients benefiting from the social security protection.

Exclusion Criteria:

* Patients under 18 years of age,
* Patients having known allergy or sensitivity to adhesive dressing materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of catheters presenting any kind of complications.. | From the insertion of the catheter to its removal, an average time frame thant can go up to 4 weeks.

SECONDARY OUTCOMES:
Number of catheter infections related to poor adherent dressings. | From the insertion of the catheter to its removal, an average time frame thant can go up to 4 weeks

OTHER OUTCOMES:
Number of participants presenting allergic adverse events | From the insertion of the catheter to its removal, an average time frame thant can go up to 4 weeks.
Costs of each dressing type strategy. | From the insertion of the catheter to its removal, an average time frame thant can go up to 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No